CLINICAL TRIAL: NCT00499915
Title: Preventing Respiratory Illness Among Premature Infants: An Asthma Education and Secondhand Smoke Reduction Study
Brief Title: NICU Asthma Education and Secondhand Smoke Reduction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Halcyon Hill Foundation (Other)
Responsible Party: Principal Investigator, Jill Halterman, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15214
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Respiratory Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secondhand Smoke Reduction and Asthma Education (Experimental): Parents of children in the experimental group will receive asthma education at NICU discharge as well as a secondhand smoke reduction program.
  Interventions: Behavioral: Secondhand Smoke Reduction and Smoking Cessation Counseling; Behavioral: Asthma Education
- Asthma Education (Active Comparator): Parents of children in the active comparator group will receive asthma education at NICU discharge.
  Interventions: Behavioral: Asthma Education

INTERVENTIONS:
Behavioral: Secondhand Smoke Reduction and Smoking Cessation Counseling — A secondhand smoke reduction program, including smoking cessation counseling (if appropriate), and feedback about the children's cotinine levels will be implemented using principles of Motivational Interviewing.
  Arms: Secondhand Smoke Reduction and Asthma Education
Behavioral: Asthma Education — Asthma education will be provided at NICU discharge.

SUMMARY:
Premature infants have a significantly increased risk for developing respiratory illnesses and asthma. Secondhand smoke (SHS) also is clearly associated with increased breathing problems in children, thus exposure to smoke makes it substantially more likely for a premature infant to develop wheezing. The overall goal of this study is to test whether comprehensive asthma education combined with a home-based secondhand smoke reduction program can reduce exposure to smoke and prevent respiratory illness among premature infants. Our hypotheses are:

* More premature infants whose families receive asthma education combined with a SHS reduction intervention will live in smoke-free environments compared to infants receiving only asthma education (control group).
* Caregivers receiving the SHS reduction program will have higher rates of quit attempts and less relapse into smoking compared to caregivers in the control group.
* Infants whose families receive the combined intervention will experience less respiratory illness compared to infants in the control group.

ELIGIBILITY:
Inclusion Criteria:

* ≤32 weeks gestation
* Planned discharge to home from the Neonatal Intensive Care Unit
* Parent or caregiver must consent to the intervention
* The first sibling discharged, for twins or infants from a multiple birth pregnancy

Exclusion Criteria:

* Inability to speak and understand English
* No access to a working phone for follow-up surveys (either at the subject's home or an easily accessible alternate home)
* Family residence outside the greater Rochester area (more than 30 miles away)
* Children in foster care or other situations in which guardian consent cannot be obtained
* The child having significant medical conditions, including serious heart disease, cystic fibrosis, or other conditions that could interfere with the assessment of respiratory-related outcome measures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S. Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Parents of children in the experimental group will receive asthma education at NICU discharge as well as secondhand smoke reduction program.
  Secondhand Smoke Reduction, Smoking Cessation: Parents of children in the experimental group will receive asthma education at NICU discharge as well as a secondhand smoke reduction program including feedback about the children's cotinine levels.
- Comparison: Parents of children in the active comparator group will receive asthma education at NICU discharge.
  Asthma Education with Secondhand Smoke Reduction: Parents of children in the active comparator group will receive asthma education at NICU discharge but no secondhand smoke reduction program will be implemented.
Period: Overall Study
Arm/Group | Treatment | Comparison
Started | 83 | 82
Completed | 68 | 76
Not Completed | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Comparison | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Gestational Age (weeks)
  Weeks | 28.7 (2.4) | 28.1 (2.5) | 28.4 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 49 | 49 | 98
Region of Enrollment [Number; unit: participants]
  United States | 83 | 82 | 165

OUTCOME MEASURES:

1. Primary Outcome: Infants Living in Smoke-free Environments.
Description: Infants living in homes with a "home smoking ban" rule
Time Frame: 5 months post baseline
Measure: Number; unit: participants
Arm/Group | Treatment | Comparison
Number analyzed (Participants) | 68 | 76
participants | 65 | 64

2. Secondary Outcome: Respiratory Morbidity Assessed Through Respiratory Symptoms as Well as Health Care Utilization for Respiratory Illnesses.
Time Frame: 2, 5, and 7-9 months post baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Only the infant participants were assessed for adverse events.
Arm/Group | Treatment | Comparison
Serious Adverse Events (participants affected / at risk) | 1/83 | 1/82
Other Adverse Events (participants affected / at risk) | 0/83 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=83) | Comparison (N=82)
Death (General disorders) | 1 (1) | 1 (1) — All infants in this study are born premature and at risk for other complications. These children passed away while enrolled in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No